CLINICAL TRIAL: NCT05449730
Title: An Investigation of the Gait Performance and Balance in Yoga Instructors
Status: Completed | Type: Observational
Sponsor: Cheng-Hsin General Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Other Study IDs: (929)111-08
Record Dates: First submitted 2022-06-24; First posted 2022-07-08 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Gait; Yoga; Balance
Keywords: Core muscle; Balance; Gait; Yoga; Symmetry; Inertial measurement units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Yoga instructor: (a) overall good health and can cooperate with orders reasonably; (b) between the ages of 25 to 60 years old; (c) no limb or leg discrepancy; (d) no history of surgery on the lower limbs or spine; (e) no history of musculoskeletal injury over the lower back in the past six months; (f)practice yoga three to six days per week and at least ten years of experience in yoga
- Healthy adult control: (a) overall good health and can cooperate with orders reasonably; (b) between the ages of 25 to 60 years old; (c) no limb or leg discrepancy; (d) no history of surgery on the lower limbs or spine; (e) no history of musculoskeletal injury over the lower back in the past six months; (f) no experience with yoga training; (g)participated in regular exercise 2 or 3 times a week

SUMMARY:
Yoga is a popular exercise and thought to be beneficial to many aspects such as mood, flexibility and balance, etc. Gait performance is a indicator of overall health and functional status. This study aims to investigate whether or not yoga instructors have a more symmetric gait pattern and better balance ability than healthy people without experience of performing Yoga. Inertial measurement units (IMUs) will be used to gather data related to gait symmetry and single leg stance balance. A comparison by four performance indexes related to gait symmetry and balance will be made to quantify the potential advantages of yoga practice.

DETAILED DESCRIPTION:
Yoga is a form of exercise with a focus on the structural alignment of the physical body. As Yoga movements involve a complex motion of core muscles and lower limb muscles, this exercise may be beneficial for gait stability. Gait performance is a sensitive indicator of overall health and functional status, and gait impairment can lead to a high risk of falling or diminished mobility. It was hypothesized that yoga instructors may have a more symmetric gait pattern and better balance ability than healthy non-yoga controls. Impact of yoga training on gait symmetry and single leg stance balance will be investigated. Twenty five yoga instructors and twenty five age/sex-matched healthy subjects will be recruited to conduct walking and static stability tests and these subjects' gait data and body movements will be measured during the experiments by attaching inertial measurement units (IMUs) to their lower limbs and trunks. Calculation of the subjects' asymmetry of swing phases during their gait cycles will be done to evaluate the gait performance. Afterwards, subjects will conduct four different one-leg stance tests. Two balance indexes will be defined and the recorded IMU data will be applied to evaluate the subjects' balance ability. Four performance indexes will then be defined to assess gait performance and single leg stance stability to quantify the potential advantages of yoga practice.

ELIGIBILITY:
[Yoga instructor]

Inclusion Criteria:

* overall good health and can cooperate with orders reasonably
* between the ages of 25 to 60 years old
* practicing three to six days per week and at least ten years of experience in yoga

Exclusion criteria

* limb or leg discrepancy
* history of surgery on the lower limbs or spine
* history of musculoskeletal injury over the lower back in the past six months

[Healthy control]

Inclusion Criteria:

* overall good health and can cooperate with orders reasonably
* between the ages of 25 to 60 years old
* participated in regular exercise 2 or 3 times a week

Exclusion criteria

* limb or leg discrepancy
* history of surgery on the lower limbs or spine
* history of musculoskeletal injury over the lower back in the past six months
* experience of Yoga practicing

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Yoga instructor: active and highly experienced Yoga instructor
  Healthy control: gender-matched healthy participants who had no experience with yoga training and participated in regular exercise 2 or 3 times a week
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Gait performance index of normal walk | within 1 month after recruitment
  asymmetric level of the swing phases calculated by IMU when performing normal walk
Gait performance index of Tandem gait with eyes open | within 1 month after recruitment
  asymmetric level of the swing phases calculated by IMU when performing Tandem gait with eyes open
Gait performance index of Tandem gait with eyes closed | within 1 month after recruitment
  asymmetric level of the swing phases calculated by IMU when performing Tandem gait with eyes closed
Open eye dominant foot standing balance indexes of chest | within 1 month after recruitment
  absolute angular velocities obtained by chest IMU when standing on the dominant foot with eyes open
Open eye dominant foot standing balance indexes of lumbar | within 1 month after recruitment
  absolute angular velocities obtained by lumbar IMU when standing on the dominant foot with eyes open
Closed eye dominant foot standing balance indexes of chest | within 1 month after recruitment
  absolute angular velocities obtained by chest IMU when standing on the dominant foot with eyes closed
Closed eye dominant foot standing balance indexes of lumbar | within 1 month after recruitment
  absolute angular velocities obtained by lumbar IMU when standing on the dominant foot with eyes closed
Open eye non-dominant foot standing balance indexes of chest | within 1 month after recruitment
  absolute angular velocities obtained by chest IMU when standing on the non-dominant foot with eyes open
Open eye non-dominant foot standing balance indexes of lumbar | within 1 month after recruitment
  absolute angular velocities obtained by lumbar IMU when standing on the non-dominant foot with eyes open
Closed eye non-dominant foot standing balance indexes of chest | within 1 month after recruitment
  absolute angular velocities obtained by chest IMU when standing on the non-dominant foot with eyes closed
Closed eye non-dominant foot standing balance indexes of lumbar | within 1 month after recruitment
  absolute angular velocities obtained by lumbar IMU when standing on the non-dominant foot with eyes closed

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Fu Chen, MD/PhD, Principal Investigator — Cheng-Hsin General Hospital
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan